CLINICAL TRIAL: NCT00893763
Title: Oral Care Intervention in Mechanically Ventilated Adults
Brief Title: Strategies To Prevent Pneumonia 2 (SToPP2)
Acronym: SToPP2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of South Florida (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2R01NR007652 (NIH); R01NR007652 (NIH)
Record Dates: First submitted 2009-05-04; First posted 2009-05-06 (Estimated); Results first posted 2016-01-11 (Estimated); Last update posted 2016-01-11 (Estimated); Status verified 2015-12

CONDITIONS: Infections, Hospital; Ventilator-Associated Pneumonia; Mechanical Ventilation Complication
Keywords: Nosocomial (Hospital-Acquired) Infections; Ventilator-Associated Pneumonia; Mechanical ventilation; Endotracheal intubation
MeSH Terms: conditions — Cross Infection; Pneumonia, Ventilator-Associated; Infections

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pre-intubation CHX (Experimental): Chlorhexidine applied to oral cavity prior to intubation
  Interventions: Procedure: Pre-intubation CHX
- Control (Active Comparator): No chlorhexidine applied to oral cavity prior to intubation
  Interventions: Procedure: Control

INTERVENTIONS:
Procedure: Pre-intubation CHX — Oral application of 5 ml CHX gluconate 0.12% solution pre-intubation, and 5 ml CHX gluconate 0.12% solution twice a day following intubation.
  Arms: Pre-intubation CHX
Procedure: Control — No pre-intubation intervention, 5 ml CHX gluconate 0.12% solution twice a day following intubation
  Arms: Control

SUMMARY:
Ventilator-associated pneumonia (VAP) is a serious complication in mechanically ventilated critically ill patients. The intervention tested in this project (swabbing the mouth with chlorhexidine before the endotracheal tube is inserted) could reduce the risk of ventilator-associated pneumonia.

DETAILED DESCRIPTION:
Ventilator-associated pneumonia (VAP) is an acute care complication with high morbidity and mortality, which is costly in length of stay and resources used. Application of chlorhexidine (CHX) to the mouths of critically ill adults after intubation reduces risk of VAP. During intubation, organisms may be dragged by the tube from the contaminated mouth to the sterile lung, and the endotracheal tube (ET) provides a pathway for direct entry of bacteria from the mouth to the lower respiratory tract. However, procedures to decontaminate the mouth before intubation are not routine and little is known about the effects of pre-intubation CHX in critically ill patients. Thus, this project focuses on evaluating the benefit of adding a pre-intubation CHX dose to the known benefit of post-intubation CHX to reduce the risk of VAP. In order to examine the effect of pre-intubation CHX on early ET colonization, we will perform microbial cultures of ETs of subjects who are extubated in the first 24 hours of study participation. We will also explore selected biomarkers (procalcitonin, cytokines) as indicators of development of VAP in a subset of subjects. The project will add to knowledge about the relationships among oral health, ET intubation and VAP, and addresses an important clinical outcome. Pre-intubation oral decontamination could reduce risk of VAP and its associated morbidity and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Need for intubation

Exclusion Criteria:

* Pneumonia at the time of intubation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 314 (Actual)
Dates: Start 2008-09; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cindy L Munro, RN,ANP,PHD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

REFERENCES:
- [Result] Munro CL, Grap MJ, Sessler CN, Elswick RK Jr, Mangar D, Karlnoski-Everall R, Cairns P. Preintubation application of oral chlorhexidine does not provide additional benefit in prevention of early-onset ventilator-associated pneumonia. Chest. 2015 Feb;147(2):328-334. doi: 10.1378/chest.14-0692. PMID 25317722

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled from two large urban teaching medical centers (VCU Health System, Tampa General Hospital). Subjects were recruited in multiple clinical areas just prior to intubation, including critical care units, emergency departments, pre-operative areas, procedural areas, and medical-surgical units during rapid response or code calls.
Groups:
- 1: Preintubation Oral Chlorhexidine: Intervention: Oral application of 5 ml CHX gluconate 0.12% solution pre-intubation, and 5 ml CHX gluconate 0.12% solution twice a day following intubation.
- 2: Control: Control: No pre-intubation intervention, 5 ml CHX gluconate 0.12% solution twice a day following intubation
Period: Overall Study
Arm/Group | 1: Preintubation Oral Chlorhexidine | 2: Control
Started | 157 | 157
Completed | 47 | 47
Not Completed | 110 | 110
Not completed — extubated | 110 | 110

BASELINE CHARACTERISTICS:
Population: Adults requiring endotracheal intubation
Groups:
- Total: Total of all reporting groups
Arm/Group | 1: Preintubation Oral Chlorhexidine | 2: Control | Total
Number analyzed (Participants) | 157 | 157 | 314
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.08 (15.85) | 58.20 (16.19) | 58.12 (16.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66 | 98 | 164
  Male | 91 | 59 | 150
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 4 | 9
  Not Hispanic or Latino | 152 | 153 | 305
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 45 | 56 | 101
  White | 106 | 96 | 202
  More than one race | 6 | 5 | 11
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 157 | 157 | 314

OUTCOME MEASURES:

1. Primary Outcome: Development of VAP (Clinical Pulmonary Infection Score)
Description: Change between post-intervention CPIS and baseline CPIS. Serial prospective evaluation of VAP risk. 6 elements of CPIS (tracheal secretions, temperature, white blood count, oxygenation, chest radiograph, and tracheal aspirate culture) summed to yield total score of 0-12 daily; higher score reflects greater likelihood of VAP.
Time Frame: Baseline up to 5 days
Population: Subjects who had complete CPIS data on admission to the study (Day 0) and subsequent complete CPIS data from day 2, 3, 4 or 5 (47 CHX & 47 control, 438 observations) were included in the analysis in accordance with intent to treat analysis principles.
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- 1: Preintubation Intervention: Intervention: Oral application of 5 ml CHX gluconate 0.12% solution pre-intubation, and 5 ml CHX gluconate 0.12% solution twice a day following intubation.
Arm/Group | 1: Preintubation Intervention | 2: COntrol
Number analyzed (Participants) | 47 | 47
units on a scale | 4.13 (0.28) | 4.45 (0.31)
Statistical Analysis 1: Comparison: 1: Preintubation Intervention vs 2: COntrol; We compared groups in a single analytical model using a mixed effects linear model with CPIS as the response variable. For this model, group (CHX, control), day, group by day interaction, APACHE III score and hospital (VCU, USF) were modeled as fixed effects and subject was modeled as a random effect; Test type: Superiority or Other; p = 0.1763, mixed effects linear model
Statistical Analysis 2: Comparison: 1: Preintubation Intervention vs 2: COntrol; A logistic regression analysis was performed using the binary response variable of colonization or no colonization and dependent variables for group, length of intubation, and group-by-length-of-intubation interaction. The probability of a type 1 error ( a ) was set to 0.05; Test type: Superiority or Other; p = 0.8656, Regression, Logistic

2. Secondary Outcome: Endotracheal Tube Colonization
Description: semiquantitative swab culture for potentially pathogenic organisms of distal end of the endotracheal tube (ETT) interior lumen at extubation. Results were collapsed into two categories: colonization (moderate or many organisms) or no colonization.
Time Frame: 24 hours
Population: The subjects analyzed were a subset of subjects enrolled in the study from whom endotracheal tunes were obtainable for microbial culture post-intubation. Subset analysis was planned a priori.
Measure: Number; unit: percentage of ET tubes colonized
Arm/Group | 1: Preintubation Oral Chlorhexidine | 2: Control
Number analyzed (Participants) | 43 | 40
percentage of ET tubes colonized | 18.6 | 17.5

3. Secondary Outcome: Serum Cytokines
Time Frame: 5 days
Reporting Status: Not Posted

4. Secondary Outcome: Serum Procalcitonin
Time Frame: 5 days
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 10 days
Description: Medical record review Medical provider report
Groups:
- 1: Intervention: Intervention: Oral application of 5 ml CHX gluconate 0.12% solution pre-intubation, and 5 ml CHX gluconate 0.12% solution twice a day following intubation.
Arm/Group | 1: Intervention | 2: Control
Serious Adverse Events (participants affected / at risk) | 0/157 | 0/157
Other Adverse Events (participants affected / at risk) | 0/157 | 0/157

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No